CLINICAL TRIAL: NCT03939351
Title: Multimodal Imaging Analysis, OCT-angiography (Optical Coherence Tomography) and SD-OCT (Spectral Domain Optical Coherence Tomography), of Retinal and Choroidal Variations Observed After a Revascularization Procedure on the Internal Carotid Artery
Brief Title: Imagery of Retinal and Choroidal Variations Observed After a Revascularization Procedure on the Internal Carotid Artery
Acronym: CAROCT-A
Status: Withdrawn | Type: Observational
Why Stopped: withdrawal of the project
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: CAROCT-A; 2018-A00777-48 (Other: ID-RCB)
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Carotid Artery Injuries
MeSH Terms: conditions — Carotid Artery Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: OCT-angiography and SD-OCT — Performing an OCT-angiography and SD-OCT examination

SUMMARY:
The purpose of this study is to describe the changes in morphology and Retinal vascularization after revascularization of the internal carotid artery. Indeed, the stenosis of the internal carotid artery can lead to ophthalmological charts. The underlying hypothesis is that revascularization of the internal carotid artery would improve ipsilateral and retinal homolateral perfusion in the short term. The OCT-angiography technique accurately studies the retinal vasculature and also assesses the risk of retinal and choroidal embolism, which is recognized as increased in cases of symptomatic or asymptomatic carotid stenosis.

DETAILED DESCRIPTION:
The stenosis of the internal carotid artery is a frequent and potentially serious pathology (TIA, ischemic stroke, death), which can also be manifested by ophthalmological charts, foremost among which are transient monocular blindness.

The most common etiology of this stenosis remains the atheromatous pathology, whose treatment, depending on the symptomatic or non-symptomatic nature of the stenosis, includes, among other things, a revascularization procedure that may be surgical (endarterectomy, reference treatment) or guided by radiology (angioplasty and carotid stent placement)

From the anatomical point of view, the internal carotid artery notably has for branching the ophthalmological artery, which itself will give birth:

* at the central artery of the retina: role in the vascularization of the inner layers of the retina
* posterior ciliary arteries: role in the choroidal vasculature and outer layers of the retina.

Very little knowledge at the present time relates changes in retinal and choroidal vascularization after a revascularization procedure on the internal carotid artery OCT-angiography is a non-invasive imaging technique that is now part of investigative examinations in retinal imaging. This technique makes it possible to study the macular and choroidal retinal vascularization with precision without injection of contrast medium and thus allows to deepen the knowledge in medical fields where the exploration was until now limited because of the invasiveness of the examinations.

The hypothesis of this project is that revascularization of the internal carotid artery would improve retinal and choroidal ipsilateral perfusion in the short term (1 month postoperatively), as assessed by OCT-angiography. OCT-angiography could also be used to assess retinal and choroidal embolism risk, usually recognized as increased in cases of symptomatic or asymptomatic carotid stenosis.

ELIGIBILITY:
Inclusion Criteria

* Patient aged 18 or over
* Indication of treatment with a carotid revascularization procedure (conventional surgery or angioplasty and stent)
* Acceptance to participate in the protocol

Exclusion Criteria:

* Associated retinal ophthalmological pathology: diabetic retinopathy, age-related macular degeneration, retinal vein occlusion, CRSC (Central serous chorioretinopathy)
* Refusal to participate in the study
* Not affiliated to a social security scheme

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be proposed to patients for whom revascularization has been performed by vascular surgeons (symptomatic, asymptomatic carotid stenosis)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
homolateral retinal and choroidal vascular density (%) | 1 month
  Finely describe the homolateral retinal and choroidal vascular density changes in the macula in OCT-angiography at 1 month after revascularization on the internal carotid artery

SECONDARY OUTCOMES:
Vascular density of contralateral eye (%) | 1 month
  Describe the variations of vascular density in OCT-A on the controlateral eye after revascularization
Subfoveal choroidal thickness | 1 month
  Describe the variations of subfoveal choroidal thickness in OCT-EDI (Enhanced depth imaging optical coherence tomography) after revascularization
Optical fiber thickness | 1 month
  Describe the variations in homolateral optical fiber thickness in RNFL ( Retinal Nerve Fiber Layer)OCT after revascularization
retinal and choroidal vascular density (%) | 1 month
  Compare the retinal and choroidal variations according to the proposed procedure: conventional surgery or angioplasty and stenting
Intraocular pressure (mm Hg) | 1 month
  Compare changes in intraocular pressure before and after revascularization procedure
Retinal and choroidal vascular density (%) according to the type of carotid stenosis | 1 month
  Compare changes in retinal and choroidal vascular density according to the type of carotid stenosis: symptomatic stenosis, asymptomatic stenosis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Henri-Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No